CLINICAL TRIAL: NCT06936891
Title: Virtual Ward for Early Discharge in Patients Receiving Inpatient Care: A Prospective Feasibility Study on Home Monitoring for the Early Discharge of Eligible Hospitalized Patients in an Outpatient Setting
Brief Title: Virtual Ward for Early Discharge in Patients Receiving Inpatient Care
Acronym: VIP care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Michael Cornelis van Herwerden, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MEC-2024-0060
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Early Discharge; Telemedicine; Virtual Clinic; Hospital at Home; Feasibility Studies
Keywords: early discharge; telemedicine; virtual ward; virtual clinic; hospital at home; feasability; telemonitoring

STUDY DESIGN:
Intervention Model Description: In this single-group study, patients eligible for early discharge are enrolled into a Virtual Ward model, providing hospital-level care at home. Care includes diagnostics (e.g., laboratory and urine testing) and treatment (e.g., intravenous antibiotics) equivalent to standard inpatient care, but administered in the home environment.
  Vital signs (oxygen saturation, respiratory rate, heart rate, blood pressure, weight, temperature) are monitored remotely three times daily via CE-marked devices and a secure mobile application (Digizorg), connected to the Zorgverlenerscockpit (Electronic Medical Record).
  Patients complete digital anamnesis questionnaires three times daily. Alerts for deviating vital signs or symptoms are handled by Virtual Ward staff, who verify measurements and escalate to the responsible physician if needed, according to predefined care pathways.
  Communication with patients and physicians follows standard clinical care protocols through (video) calls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Ward arm (Experimental): Patients receive hospital-level care at home via a Virtual Ward, including remote monitoring of vital signs, digital anamnesis questionnaires, and standard diagnostics and treatment, supported by telemonitoring staff and hospital physicians.
  Interventions: Combination Product: Virtual Ward

INTERVENTIONS:
Combination Product: Virtual Ward — Hospital-level care at home using remote vital sign monitoring, digital anamnesis via the Digizorg app, and integration with the Electronic Medical Record (HiX), managed by Virtual Ward staff following predefined care pathways.

SUMMARY:
This study evaluates the feasibility of providing hospital-level care at home for eligible patients through a Virtual Ward. Patients are discharged early from the hospital and monitored remotely using digital vital sign monitoring and anamnesis questionnaires. The primary aim is to determine if at least 30% of eligible patients can be safely and successfully transferred to the Virtual Ward under current Dutch healthcare conditions.

DETAILED DESCRIPTION:
Rationale: Patients undergo extensive diagnostics and treatment adjustments during the early days of their hospitalization, which may become less imperative as their admission progresses. If a patient's vital signs stabilize after the initial hospitalization, and they only necessitate "less urgent" hospital care, an option is to transfer them to the Virtual Ward and thereby creating hospital capacity. This telemedicine-driven model presents an alternative to the conventional in-patient care approach. In the Virtual Ward, patients continue to receive care under supervision of the hospital physician but from the comfort of their own homes. This means the hospital oversees the monitoring of vital signs, performing diagnostics and treatment in the patient's home environment. A growing body of evidence supports the safety of "Virtual Wards." However, although proven safe, its feasibility remains uncertain.

Objective: To assess the feasibility of the Virtual Ward in six pre-defined sub-cohorts of non elective hospitalized patients within the current Dutch healthcare system.

Study design: This is a single-center prospective cohort trial with 6 sub-cohorts.

Study population: Admitted patients (minimum age 18) receiving inpatient care that are eligible for discharge to the Virtual Ward.

Intervention (if applicable): Patients will be discharged to the Virtual Ward with monitoring, diagnostics, and treatment at home.

Main study parameters/endpoints: To assess the feasibility of the Virtual Ward across six pre-defined sub-cohorts of non-elective hospitalized patients by determining the percentage of patients who provide informed consent and are successfully transferred to the Virtual Ward, with a feasibility threshold set at 30% for this pilot phase (adherence). Feasibility is determined per sub-cohort.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients who are admitted to the virtual ward can benefit from recovering in a home environment. Potential risks are that they are not within reach of the treating physicians in case of an adverse event. Patients need to fill in questionnaires and measure their own vital signs. There are no additional invasive interventions patients would need to undergo by participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old).
* Currently hospitalized and eligible for early discharge according to clinical judgment.
* Ability to provide written informed consent.
* Access to a smartphone or tablet with internet connection.
* Patient is capable of using the Digizorg app or has support from a caregiver who can assist.
* Suitable home situation for Virtual Ward care (e.g., safe environment, necessary utilities available).
* Enrollment in one of the predefined Virtual Ward care pathways

Exclusion Criteria:

* Patients requiring continuous hospital-based monitoring or interventions that cannot be safely delivered at home.
* Patients who are hemodynamically unstable or require oxygen therapy >5 liters/minute at the time of discharge.
* Patients unable or unwilling to comply with home monitoring procedures.
* Patients with significant cognitive impairment without adequate caregiver support.
* Patients with a life expectancy less than 30 days, as assessed by the treating physician.
* Patients participating in another interventional clinical trial that could interfere with the Virtual Ward protocol.
* Any other condition that, in the opinion of the treating physician, would make participation unsafe or infeasible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Successfully Transferred to the Virtual Ward After Providing Informed Consent | From enrollment to transfer to Virtual Ward (during hospitalization, up to 7 days)
  Successful transfer is defined as discharge from hospital to the Virtual Ward with start of home monitoring according to care pathways. Threshold for feasibility is ≥30%.

SECONDARY OUTCOMES:
Number of Eligible Patients Invited for Participation | From enrollment to invitation during hospitalization (up to 7 days)
  Eligible patients are those meeting the inclusion criteria, identified during hospitalization.
Number of Invited Patients Providing Informed Consent | From enrollment to signing informed consent during hospitalization (up to 7 days)
  Informed consent is obtained after providing oral and written information.
Time from Study Inclusion to Transfer to Virtual Ward | From informed consent to Virtual Ward admission (up to 7 days)
  Time is measured in days between signing informed consent and actual discharge to Virtual Ward.
Number of Notifications Generated During Virtual Ward Monitoring | From Virtual Ward admission up to 30 days after discharge
  Notifications include vital sign alerts or digital anamnesis alerts, categorized into low-exceeding or high-exceeding limits.
Number of Contact Moments with Virtual Ward Staff | From Virtual Ward admission up to 30 days after discharge
  Contact moments include staff-initiated, patient-initiated, and home nurse-initiated contacts recorded with reasons.
Length of Stay in Hospital Ward Prior to Virtual Ward Transfer | From hospital admission to Virtual Ward admission
  Measured in days from hospital admission to discharge to the Virtual Ward
Length of Stay in the Virtual Ward | During Virtual Ward stay
  Measured in days from Virtual Ward admission to discharge from Virtual Ward.
Hospital Readmission Rate During Virtual Ward Stay | During Virtual Ward stay
  Readmission is defined as return to hospital ward due to clinical deterioration or treatment need.
Hospital Readmission Rate Within 30 Days After Virtual Ward Discharge | From Virtual Ward discharge up to 30 days
  Readmission defined as hospitalization for clinical reasons after Virtual Ward discharge.
Change in Quality of Life as Measured by EQ-5D-3L | From baseline (hospital inclusion) to end of Virtual Ward treatment
  EQ-5D-3L score ranges from 0 (worst health) to 1 (best health). Difference between baseline and end of Virtual Ward stay will be measured.

OTHER OUTCOMES:
Frailty Status Based on Clinical Frailty Scale and PRISMA-7 Questionnaire | At enrollment (baseline)
  Clinical Frailty Scale: 1 (very fit) to 9 (terminally ill); PRISMA-7 score: ≥3 indicates frailty risk.
Patient-Reported Experience of Virtual Ward Care | Within 30 days after Virtual Ward discharge
  Semi-structured interview assessing experiences, barriers, and facilitators, based on CFIR.
Healthcare Provider-Reported Experience of Virtual Ward Care | Approximately 6-12 months after study initiation
  Semi-structured interview assessing experiences using CFIR domains and NoMAD questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Cox van de Weg, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided